CLINICAL TRIAL: NCT05918770
Title: Telemedicine-guided Patients Reported Outcome Measures (PROMs): Side Effects Screening and Early Intervention to Impact in Quality of Life of Gynaecological Cancer Patients
Brief Title: Side Effects Screening and Early Intervention to Impact in Quality of Life of Gynaecological Cancer Patients
Acronym: HALIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Blanca Gil Ibañez, Principal Investigador, MD, PhD, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nº CEIm: 23/157
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life; Gynaecological Cancer; Lymphedema, Lower Limb; Sexual Dysfunction
Keywords: quality of life; Gynaecological cancer
MeSH Terms: conditions — Lymphedema; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): in case of positive screening, the online app will alert and the patient will be referred to the corresponding area for diagnosis and early treatment (Rehabilitation, Psycho-oncology, Sexual health and Nutrition)
  Interventions: Diagnostic Test: systematic screening and early treatment
- control group (No Intervention): will follow the standard usual care guidelines at the centre where patients will be opportunistically referred to specialised care

INTERVENTIONS:
Diagnostic Test: systematic screening and early treatment — in case of positive screening, the online app will alert and the patient will be referred to the corresponding area for diagnosis and early treatment (Rehabilitation, Psycho-oncology, Sexual health and Nutrition
  Arms: experimental group

SUMMARY:
The goal of this randomized study is to assess the impact on self-perceived quality of life (QoL) of systematic screening and early treatment of aftereffects in patients with gynaecological cancers. The main question it aims to answer is if systematic screening with validated questionaries (see in detailed description), diagnosis and early treatment of lower-limb lymphoedema, anxiety-depression, sexual dysfunction and sarcopenia-malnutrition all have a positive impact on the self-perceived QoL by gynaecological cancer patients. Participants will access the screening questionnaires and QoL questionaries on a free online app on their mobile devices. In the experimental group, in case of positive screening, patients will be referred to specialised care to early treatment of the aftereffects. Researchers will compare this group with standard usual care (opportunistic treatment) to see if systematic screening and early treatment lead to a better QoL.

DETAILED DESCRIPTION:
validated screening scales used: Gynecologic Cancer Lymphedema Questionnaire (GCLQ) Hospital Anxiety and Depression Scale (HADS) Sexual Function Abbreviated Index (IFSFA-6) Short Nutritional Assessment Questionnaire (SNAQ) Sarcopenia Formulary (SARC-F) along with self-perceived quality of life questionnaires from EORTC: QLQ-C30 EN-24 or OV-28 or CX-24

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 diagnosed with ovarian, tubal and primary peritoneal, cervical and endometrial cancer who are candidates for surgery during the study period.

Exclusion Criteria:

* Patients unable to complete by themselves the screening questionnaires included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life questionaries score | up to 20 months
  Unit on QLQ-C30 Quality-of-life scale

SECONDARY OUTCOMES:
Quality-of-life questionaries score related to endometrial cancer | up to 20 months
  Unit on QLQ-EN-24 Quality-of-life scale
Quality-of-life questionaries score related to cervical cancer | up to 20 months
  Unit on QLQ-Cx-24 Quality-of-life scale
Quality-of-life questionaries score related to ovarian cancer | up to 20 months
  Unit on QLQ-Ov-28 Quality-of-life scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gil-Ibanez B, Tejerizo-Garcia A, Oliver MR, Madariaga A, Maiz Jimenez M, Gil Garcia A, Lopez-Gonzalez G. Side effects screening and early intervention to impact in quality of life of patients with gynecological cancers (HALIS study). Int J Gynecol Cancer. 2023 Oct 2;33(10):1645-1648. doi: 10.1136/ijgc-2023-004802. PMID 37748803